CLINICAL TRIAL: NCT06877520
Title: Early Feasibility Study (EFS) of the 'Pivot Extend' in Treatment for Tricuspid Regurgitation (SPACER Study)
Brief Title: Early Feasibility of 'Pivot Extend' for Tricuspid Regurgitation Treatment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tau-MEDICAL Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TCP-EFS-07-GE
Record Dates: First submitted 2025-03-10; First posted 2025-03-14 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Tricuspid Regurgitation (TR)
Keywords: Pivot Extend; TauMedical
MeSH Terms: conditions — Tricuspid Valve Insufficiency

STUDY DESIGN:
Intervention Model Description: Multi-center, open label, single arm, early feasibility study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment to Improve TR Symptoms with Investigational Medical Device Implantation (Experimental): Participants assigned to this arm will receive an investigational medical device designed to improve symptoms of severe and clinically symptomatic tricuspid regurgitation (TR). Following device implantation, participants will be monitored in a specialized facility for at least 24 hours with real-time observation of vital signs. The device's safety and efficacy will be assessed over 12 months through scheduled visits, with clinical progress monitored throughout. Device removal may be performed if adverse events occur or if deemed necessary by the investigator.
  Interventions: Device: Pivot Extend Tricuspid Regurgitation Spacer Device

INTERVENTIONS:
Device: Pivot Extend Tricuspid Regurgitation Spacer Device — The Pivot Extend Tricuspid Regurgitation Spacer Device is an investigational implant designed to reduce tricuspid regurgitation (TR) by occupying the regurgitant orifice and improving leaflet coaptation. The device is implanted via a transcatheter procedure under imaging guidance. Following implantation, participants will undergo post-procedural monitoring for at least 24 hours to ensure safety and device stability. The device is intended for long-term placement, with scheduled follow-up assessments at designated intervals over a 12-month period to evaluate its safety and efficacy. Device removal may be performed if adverse events occur or if deemed necessary by the investigator.

SUMMARY:
This clinical trial aims to evaluate the safety and demonstrate the efficacy of treatment to improve tricuspid regurgitation (TR) symptoms in patients with severe and clinically symptomatic TR through long-term implantation of an investigational medical device.

1. Determine the safety of long-term implantation of the investigational medical device "Pivot Extend" by monitoring for MACEs associated with the investigational medical device or procedure that may occur with long-term associated with the investigational medical device or procedure that may occur with long-term implantation.
2. Device success, procedural success, and clinical outcomes of long-term implantation of the investigational medical device "Pivot Extend" will be monitored.

ELIGIBILITY:
Inclusion Criteria:

1. Adults 18 years of age or older at the time of screening
2. Those with symptoms despite medical therapy (OMT, diuretics/medications) for TR for at least 1 month at screening
3. Those who meet the criteria of severe (3+) or worse on the TR grade classification table on echocardiography performed at the screening visit
4. Those with clinical symptoms of New York Heart Association (NYHA) class 2 or worse
5. Those deemed suitable for percutaneous valve intervention by a Heart Team that includes at least one cardiologist, one cardiac surgeon and one anesthesiologist.
6. Those who have voluntarily decided to participate in this clinical trial and have provided written informed consent
7. Those who can understand and follow the investigator's instructions and are able to participate for the entire duration of the study

Exclusion Criteria:

1. Those with blood clots, emboli, masses, or growths in the vascular system of the heart or lungs on an echocardiogram and cardiac CT scan performed at the screening visit
2. Those with uncorrected blood clotting disorders based on hemanalysis performed at the screening visit
3. Those who are unable to use anticoagulant agents (NOAC ex.Xarelto)
4. Those who have had major bleeding (not including minor bleeding, such as a nosebleed that can be hemostasized) treated with anticoagulants prior to participation in this clinical trial
5. Those with severe anemia (hemoglobin ≦10g/dL) that requires hospitalization
6. Those who have an implanted device such as an implantable cardioverter defibrillator (ICD) or pacemaker prior to participation in this clinical trial
7. Those whose anatomy, in the opinion of the investigator, is not suitable for implantation of an investigational medical device based on echocardiogram and cardiac CT scan performed at the screening visit
8. Those who require surgery or interventional procedures (coronary artery bypass graft (CABG) or surgery for atrial septal defect (ASD)) based on an echocardiogram performed at the screening visit
9. Those with a platelet count of 80,000/uL or less based on hemanalysis performed at the screening visit
10. Patients with pulmonary arterial hypertension with a TR Vmax greater than 3.5 m/s on echocardiography performed at the screening visit or a pulmonary vascular resistance of more than 3 Wood Units on right heart catheterization
11. Those with a left ventricular ejection fraction (LVEF) of less than 50% on echocardiogram performed at the screening visit
12. Those who have had active gastrointestinal bleeding or a digestive procedure within 3 months prior to participation in this study (those with the potential for gastrointestinal bleeding)
13. Those with a history of cerebrovascular accident (CVA) or transient ischemic attacks (TIA) within 30 days prior to participation in this clinical trial
14. Those with a history of myocardial infarction (MI) within 30 days prior to participation in this study
15. Those with active endocarditis requiring antibiotic treatment
16. Those with malignancies with end-stage renal failure requiring hemodialysis and other chronic conditions who have a life expectancy of less than one year
17. Those with moderate or severe aortic, pulmonary artery, or mitral stenosis on echocardiogram performed at the screening visit
18. Those with moderate or worse mitral valve regurgitation or severe aortic valve regurgitation on the echocardiogram performed at the screening visit
19. Those with calcification of the tricuspid valve lobes affecting the procedure on an echocardiogram performed at the screening visit
20. Those who have participated in another clinical trial within 30 days prior to participation in this clinical trial
21. Pregnant or nursing women, or women planning to become pregnant during the clinical trial period
22. Women of childbearing potential who are not using a medically accepted birth control method
23. Those with a coexisting condition, which most likely limits the participant´s life expectancy to less than one year.
24. Those with a preexisting pulmonary valve prosthesis or RV to PA conduit.
25. Those with clinical findings other than the above that, in the opinion of the investigator, are medically inappropriate for this clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Major Adverse Cardiac Events(MACEs) | 1 month post-procedure
  Occurrence Ratio of Major Adverse Cardiac Events (MACEs)

SECONDARY OUTCOMES:
Device Success | during procedure
  The rate of the device successfully placed at target location
Procedural Success(1) | 1-month, 6-month, 12-month post-procedure
  Changes in TR Grade: The number of the participants who had at least 1 TR grade drop, confirmed through echocardiography
Procedural Success(2) | 1-month, 6-month, 12-month post-procedure
  The occurrence rate of MACEs associated with the trial device or procedure
Clinical Outcomes(1) | 6-month, 12-month post-procedure
  Changes in anatomical structure: Changes in right ventricular volume from baseline confirmed through cardiac CT
Clinical Outcomes(2) | 1-month, 6-month, 12-month post-procedure
  Changes in NHYA Functional Class: The number of participants whose NYHA functional class improved compared to baseline
Clinical Outcomes(3) | 1-month, 6-month, 12-month post-procedure
  Changes in Six Minute Walk Test (6MWT): Changes in distance compared to baseline
Clinical Outcomes(4) | 1-month, 6-month, 12-month post-procedure
  Changes in KCCQ score: Changes in the assessed KCCQ score compared to baseline
Clinical Outcomes(5) | 1-month, 6-month, 12-month post-procedure
  Changes in edema score: The number of participants who had at least 1 level improvement in edema score compared to baseline
Clinical Outcomes(6) | 1-month, 6-month, 12-month post-procedure
  Changes in eGFR (estimated glomerular filtration rate): Changes in eGFR compared to baseline

CONTACTS AND LOCATIONS:
Locations (3):
- Georgia (3):
  - Israeli-Georgian Medical Research Clinic Healthycore, Tbilisi, K'alak'i T'bilisi
  - Tbilisi Heart and Vascular Clinic, Tbilisi, K'alak'i T'bilisi
  - Tbilisi Heart Center, Tbilisi, K'alak'i T'bilisi